CLINICAL TRIAL: NCT04035044
Title: Study of the Analytical Performance of ALLEGRO™ Instrument: Performance Evaluation of In Vitro Diagnostic Device
Brief Title: Study of the Analytical Performance of ALLEGRO™ Instrument
Status: Completed | Type: Observational
Sponsor: Nova Biomedical (Industry)
Collaborators: C-TRIC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 225107
Record Dates: First submitted 2019-03-13; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A new analyser has been developed (Allegro™) which allows the tests to be undertaken at the clinic, with the results available in a few minutes. This means that patients can get immediate feedback and that the doctors/nurses can adjust treatment before the patient leaves the clinic. It is obviously important that this analyser performs to a similar degree of accuracy to the laboratory analyses.

DETAILED DESCRIPTION:
Blood and urine tests are used in the assessment of diabetes and to guide clinical management. In the traditional model of care, blood samples are taken from patients at the clinic and are sent to the laboratory for analysis and the results may not be available for a number of hours/days after the clinic visit.

A new analyser has been developed (Allegro™) which allows the tests to be undertaken at the clinic, with the results available in a few minutes. This means that patients can get immediate feedback and that the doctors/nurses can adjust treatment before the patient leaves the clinic. It is obviously important that this analyser performs to a similar degree of accuracy to the laboratory analyses.

The aim of this research study is to assess the accuracy of the Allegro™ analyser compared to laboratory analyses on finger prick capillary blood samples and urine samples. Fifty (50) patients with diabetes will be invited to give a venous blood sample, finger prick capillary blood sample and urine sample. The venous blood sample, finger prick capillary blood sample and urine sample will be analysed by both the Allegro™ analyser and laboratory analyses and the results compared. The Allegro™ results will not be used in the management of the patients' diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes patients attending Altnagelvin Area Hospital Clinics or primary care in Western Trust area aged 18-80 years of age

Exclusion Criteria:

* Patients who are less than 18 years or over 80 years of age

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Fifty(50) patients with diabetes will be recruited from Diabetes Clinics, WHSCT or from patients attending primary care diabetes services.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Analytical verification of Allegro - HbA1c comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for HbA1c blood results in mmol/mol
Analytical verification of Allegro - Cholesterol comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Cholesterol blood results in mmol/L
Analytical verification of Allegro - HDL comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for HDL blood results in mmol/L
Analytical verification of Allegro - Triglycerides comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Triglycerides blood results in mmol/L
Analytical verification of Allegro - Glucose comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Glucose blood results in mmol/L
Analytical verification of Allegro - Creatinine comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Creatinine blood results in mg/dL
Analytical verification of Allegro - Urine creatinine comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Creatinine urine results in mg/dL
Analytical verification of Allegro - Urine Albumin comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Albumin urine results in g/L

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Milojkovic, PhD, Study Director — Nova Biomedical
Locations (1):
- C-TRIC, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

DOCUMENTS (1):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT04035044/Prot_000.pdf